CLINICAL TRIAL: NCT04420286
Title: Study of the Increase in ICU Beds Capacity and Caregivers During COVID-19 Pandemic in France : the FRENCH ICU Study
Brief Title: Study of the Increase in ICU Beds Capacity During COVID-19 Pandemic in France
Acronym: FRENCH ICU
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: 30RC20_0117
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2021-08

CONDITIONS: Coronavirus Infections; COVID19 Outbreak in France
Keywords: COVID-19; Critical care; Intensive Care
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hospital having ICU beds: Hospital having ICU beds during COVID-19 outbreak in France

SUMMARY:
For preventing the overwhelming of ICU beds capacity during COVID-19 pandemic in France, national and regional Health-Care institutions decided to optimize the Intensive Care Unit beds availability by opening new ICU beds in institutions with and without prior ICU. The Present study was design to retrospectively describe the origin of the ICU beds and human resources created during the COVID-19 outbreak in France.

DETAILED DESCRIPTION:
Since December 2019, the SARS-CoV-2 coronavirus disease has caused a worldwide outbreak of respiratory illness that rapidly invaded leading the world (WHO). Its most severe form is dominated by an acute respiratory distress syndrome (ARDS) with other organ failures requiring mechanical ventilation and admission in Intensive Care Unit (ICU). With a wide pandemic effect and a long length of mechanical ventilation, the intensive care units were quickly full.

For preventing the overwhelming of ICU beds capacity, national and regional Health-Care institutions (then French Health minister, every Regional Health) decided to optimize the Intensive Care Unit beds availability by opening new ICU beds in institutions with and without prior ICU.

Daily ICU beds availability was assessed in each institution, and at the regional level to organize potential patient transfers across regional and national hospital. Moreover, an extraordinary mobilization and joint efforts of medical, paramedical and administrative staff allowed getting the caregivers for managing the most severe patients in each ICU. All physicians who could manage ICU patients were involved in this crisis. In this context, anesthesiologists (who have gotten an ICU education during their studies) were involved, as the surgical activity has been reduced to the vital procedures. This overall organization permitted the admission of more patients than the initial maximum national capacity of ICU beds.

ELIGIBILITY:
Inclusion Criteria:

* Hospital having ICU during COVID-19 outbreak in France

Exclusion Criteria:

* Hospital refuse to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study is not based on patients but on hospital organisation to describe the origin of the ICU beds and human resources created during the COVID-19 outbreak in France.
Sampling Method: Non-Probability Sample
Enrollment: 9860 (Actual)
Dates: Start 2020-05-06 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
origin of the ICU beds created during the COVID-19 outbreak in France. | DAY 0
  Describe the origin of the ICU beds created during the COVID-19 outbreak in France.

SECONDARY OUTCOMES:
Human Resources | DAY 0
  Describe the human resources (medical and non-medical) mobilized to ensure that all acute patients could be managed (physicians according to their initial specialty, nurses and nursing auxiliaries).

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nîmes, Hôpital Universitaire Carémeau, Nîmes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lefrant JY, Fischer MO, Potier H, Degryse C, Jaber S, Muller L, Pottecher J, Charboneau H, Meaudre E, Lanot P, Bruckert V, Plaud B, Dureuil B, Samain E, Bouaziz H, Ecoffey C, Capdevila X; French ICU study investigators group. A national healthcare response to intensive care bed requirements during the COVID-19 outbreak in France. Anaesth Crit Care Pain Med. 2020 Dec;39(6):709-715. doi: 10.1016/j.accpm.2020.09.007. Epub 2020 Oct 5. PMID 33031979